CLINICAL TRIAL: NCT00126347
Title: Effect of Lowering of Plasma Homocysteine Concentrations After an Oral Methionine Load on Vascular Function in Healthy Volunteers
Brief Title: Effect of Betaine, Serine and Folic Acid on Vascular Function in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen Centre for Food Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: P02.0470L
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2005-08-18 (Estimated); Status verified 2005-08

CONDITIONS: Healthy; Cardiovascular Diseases
Keywords: betaine; serine; folic acid; methionine load; homocysteine; cardiovascular health; vascular function; human
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements; Betaine; Serine; Folic Acid

INTERVENTIONS:
Procedure: supplementation with betaine, serine, and folic acid

SUMMARY:
The purpose of this study is to determine whether reducing the increase in plasma homocysteine concentrations following an oral methionine load affects vascular function in healthy volunteers, irrespective of the homocysteine-lowering agent.

DETAILED DESCRIPTION:
A high plasma homocysteine is a potential risk factor for cardiovascular disease and death. However, it remains uncertain whether homocysteine per se, low status of folate, or other factors related to methionine metabolism are involved in the pathogenesis of cardiovascular disease. Previous studies have shown that a high concentration of homocysteine in blood is related to an impaired vascular function in the arteries, an indicator of cardiovascular disease risk. Virtually all intervention trials used folic acid as a homocysteine-lowering agent, which may however affect vascular function through mechanisms not related to homocysteine. The researchers investigated whether reduction in homocysteine concentrations following a methionine load, via supplementation with serine, betaine or folic acid improves vascular function in healthy volunteers, in order to distinguish between effects of folic acid and of homocysteine-lowering per se.

Comparison: The effects of supplementation with serine, folic acid and betaine (all together with an oral methionine load) were compared to the effects of a placebo (together with a methionine load) on plasma homocysteine concentrations and on vascular function following methionine loading in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* Women postmenopausal: two or more years after last menstruation. If the uterus was surgically removed, the women must be 55 years or older
* Normal blood values for: hematology, total homocysteine, lipids, vitamin B6, vitamin B12, folic acid, liver enzymes, creatinine
* Absence of protein and glucose in urine sample
* Body mass index (BMI) between 18 and 30 kg/m2
* Good ultrasound visibility of the brachial artery, judged by a sonographer.
* Willing not to use supplements containing B-vitamins, antioxidant vitamins (A, beta-carotene, C and E) or n-3 fatty acids/fish oil supplements from screening day (>2 months before start of the study) until end of study
* Willing not to be blood or plasmapherese donor from 4 weeks before the screening day, and 4 weeks before the start of the study until the end of study

Exclusion Criteria:

* Any chronic or acute disease (e.g. diabetes, renal disease, inflammation)
* Current, or history of cardiovascular disease
* Hypertension
* Medical history or surgical events know to interfere with the study
* Fasting plasma total homocysteine > 26 micromol/L
* Alcohol consumption: women >21 consumptions/week; men >28 consumptions/week
* Weight loss or gain > 2 kg in the month prior to screening
* Any special diet (prescribed, slimming, macrobiotic or total vegetarian. Sole exclusion of meat and fish from a otherwise 'normal' western diet is allowed).
* Lactose intolerance
* Use of supplements containing B-vitamins more than once weekly in the period from 3 months before the screening day
* Participation in any other trial up to 3 months before this study
* Use of medication known to interfere with the study outcome.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-08; Study Completion 2003-07

PRIMARY OUTCOMES:
concentrations of plasma homocysteine before and following an oral methionine load
vascular function, measured as flow mediated vasodilation before and following an oral methionine load

SECONDARY OUTCOMES:
B-vitamins
blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Petra Verhoef, PhD, Study Chair — Wageningen Centre for Food Sciences
Locations (1):
- Wageningen Centre for Food Sciences, Wageningen, Netherlands